CLINICAL TRIAL: NCT01874951
Title: Randomized, Proof-Of-Concept Trial of Augmentation of Antidepressants by Low Dose Naltrexone (LDN) for Patients With Breakthrough Symptoms of Major Depressive Disorder on Antidepressant Therapy
Brief Title: Low-Dose Naltrexone (LDN) for Depression Relapse and Recurrence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston Clinical Trials (Other)
Responsible Party: Principal Investigator, David Mischoulon, MD, Staff Psychiatrist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013P000371
Record Dates: First submitted 2013-05-20; First posted 2013-06-11 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Major Depressive Disorder; Depression, Unipolar; Recurrence; Relapse
Keywords: Depression; Recurrence; Relapse; Antidepressants; Naltrexone; Drug augmentation
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Recurrence; Depression | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): In this arm, patients will receive placebo for three weeks.
  Interventions: Drug: Placebo
- Naltrexone (Experimental): In this arm, patients will receive low dose naltrexone for three weeks.
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — 1 mg of naltrexone will be given twice daily to all patients assigned to active drug.
  Other Names: LDN
  Arms: Naltrexone
Drug: Placebo — Placebo identical in appearance to naltrexone will be given twice daily to all patients assigned to placebo.
  Arms: Placebo

SUMMARY:
The purpose of this pilot study is to determine if taking a low dose of naltrexone in addition to an antidepressant medication can help treat relapse or recurrence in people with Major Depressive Disorder (MDD). The U.S. Food and Drug Administration (FDA) has approved naltrexone for the treatment of alcohol dependence and opioid dependence, but the FDA has not approved naltrexone to treat depression. The investigators hypothesize that patients with breakthrough depression on an antidepressant regimen containing a pro-dopaminergic agent assigned to treatment with low dose naltrexone will demonstrate higher rates of response compared to those patients taking placebo.

DETAILED DESCRIPTION:
We carried out a pilot double-blind, randomized, controlled study of low-dose naltrexone (LDN) 1 mg b.i.d. versus placebo augmentation in MDD patients who relapsed on dopaminergic agents. The primary aim was to test the hypothesis that patients experiencing depressive breakthrough would demonstrate greater improvement in their depression when supplementing their current antidepressant regimen with LDN versus placebo, with no significant difference in side effects.

Boston area men and women with MDD were recruited from 01/13/2014-11/11/2014 via Institutional Review Board (IRB)-approved newspaper, television, internet, and radio ads initiated by Massachusetts General Hospital (MGH) and Boston Clinical Trials (BCT). Screened and eligible patients returned one week later for a baseline visit and were randomized consecutively to double-blind treatment with placebo or LDN 1 mg b.i.d. The randomization list was generated by an online randomization program and maintained by the research pharmacist. Subjects were treated for 3 weeks, with weekly assessments. All subjects were required to continue on their baseline antidepressant regimen without changes for the duration of the study; they were likewise asked not to modify any other allowed baseline medications that they had been taking prior to entering the study. Adherence was determined by weekly pill counts; protocol violation was defined as less than 80% adherence.

Side effects were assessed at every visit using the Systematic Assessment for Treatment Emergent Effects-Specific Inquiry (SAFTEE-SI) scale (Levine and Schooler, 1992) and categorized by severity as: 0-none, 1-mild, 2-moderate, 3-severe. Because some SAFTEE items could be present at baseline, particularly in a sample of subjects taking antidepressants that could themselves produce side effects, we defined as treatment-emergent any SAFTEE side effect for which severity increased by two or more levels (e.g. from none to moderate or from mild to severe) from baseline (Mischoulon et al., 2014). Frequency of side effect was based on the number of patients reporting the side effect at any time during the study.

Suicidal ideation was assessed at each visit using the Hamilton Depression Rating Scale (HAM-D). Subjects considered to be at high risk for suicide were discontinued and referred for further evaluation and hospitalization if clinically indicated. Subjects were also discontinued for any emergence of hypomania, mania, or psychosis; a Clinical Global Improvement (CGI-I) score greater than 5 (e.g., score of 6 or 7); evidence of illicit drug use or problematic alcohol use.

At the end of the double-blind study, both responders and non-responders who completed the double-blind phase had the option of receiving open-label adjunctive treatment with LDN for 3 more weeks.

Paired and independent samples t-tests and their nonparametric counterparts (Wilcoxon's signed ranks and Mann-Whitney U tests) were used to examine and compare outcomes for each treatment arm. All analyses were two-tailed. Response and remission rates, and emergence of side effects were compared by Fisher's exact test. Effect sizes (ES) were calculated by Cohen's d (Cohen, 1988), for between-subjects comparisons (changes in depression scales from baseline to end for LDN vs. placebo) and for within-subjects comparisons (changes in depression scales from baseline to end for each separate treatment group). Correlation coefficients were calculated for use in within-subjects comparisons. Statistical analyses were carried out using SPSS version 17.0 (SPSS Inc, Chicago, Illinois).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65.
* Written informed consent.
* Meet Diagnostic and Statistical Manual (DSM-IV) criteria by Structured Clinical Interview for DSM-IV (SCID-I/P) for Major Depressive Disorder (MDD), current.
* Quick Inventory of Depressive Symptomatology - Self-Rated (QIDS-SR) score of at least 12 at both screen and baseline visits.
* Received treatment with either an Selective serotonin re-uptake inhibitors (SSRI) in combination with a dopaminergic agent, or with an antidepressant with a dopaminergic mechanism of action in adequate doses, achieved remission per American College of Neuropsychopharmacology (ACNP) Task Force guidelines for ≥3 months, currently in relapse or recurrence without dose change for at least the past 4 weeks, based on meeting DSM-IV criteria for MDD.

  1. Dopaminergic agents here include classical stimulants from the amphetamine or methylphenidate families; dopamine agonists (e.g. pramipexole); or dopamine active antidepressants like bupropion.
  2. Additionally, low dose (< 2.5 mg) Abilify, a D2 partial agonist, is believed to exert pro-dopaminergic effects and will therefore be included as a dopamine agent.
  3. Sertraline, although classified as an SSRI, has dopamine reuptake inhibiting properties believed to be relevant at higher doses (> 150 mg of sertraline), and will also therefore be considered a dopaminergic antidepressant at dose range above.
  4. Based on the finding that the norepinephrine transporter is the reuptake inhibitor for dopamine in the prefrontal cortex and the robust sustained clinical response of a patient on duloxetine and low dose naltrexone, we include duloxetine, traditionally classed as an SNRI, among the dopamine acting antidepressants.)
* During the baseline visit, patients must be on a stable dose of antidepressant regimen for the past 4 weeks.

Exclusion Criteria:

* Pregnant women or women of child bearing potential who are not using a medically accepted means of contraception (to include oral contraceptive or implant, condom, diaphragm, spermicide, intrauterine device, tubal ligation, or partner with vasectomy).
* Patients who no longer meet DSM-IV criteria for MDD during the baseline visit.
* Patients who demonstrate a greater than 25% decrease in depressive symptoms as reflected by the QIDS-SR total score - screen to baseline.
* Serious suicide or homicide risk, as assessed by evaluating clinician.
* Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease.
* Substance use disorders active within the last six months, any bipolar disorder (current or past), any psychotic disorder (current or past).
* History of a seizure disorder or clinical evidence of untreated hypothyroidism.
* Patients requiring excluded medications (including but not limited to chronic or episodic use of anorexiants, episodic hormones, episodic benzodiazepines, episodic insulin, episodic and other episodic psychotropic medications).
* Psychotic features in the current episode or a history of psychotic features, as assessed by SCID.
* History of naltrexone intolerance at any dose.
* Patients with a history of antidepressant-induced hypomania.
* Inadequate exposure time or dose of current SSRI or Serotonin-norepinephrine reuptake inhibitor (SNRI); failure to comply with at least 80% of doses.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Mischoulon, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital; Depression Research and Clinical Program, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mischoulon D, Hylek L, Yeung AS, Clain AJ, Baer L, Cusin C, Ionescu DF, Alpert JE, Soskin DP, Fava M. Randomized, proof-of-concept trial of low dose naltrexone for patients with breakthrough symptoms of major depressive disorder on antidepressants. J Affect Disord. 2017 Jan 15;208:6-14. doi: 10.1016/j.jad.2016.08.029. Epub 2016 Oct 1. PMID 27736689

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After approval by our Institutional Review Board (IRB), written informed consent was obtained. Boston area men and women with major depressive disorder (MDD) were recruited from 01/13/2014-11/11/2014 via IRB-approved newspaper, television, internet, and radio ads initiated by Massachusetts General Hospital (MGH) and Boston Clinical Trials (BCT).
Pre-assignment Details: 21 prospective subjects were screened. The following were excluded: sub-threshold Hamilton-D (HAMD) scores (n=3); too recent changes in medication regimen (n=2); cerebrovascular accident in past 5 years (n=1); no history of past treatment response (n=1); inappropriate antidepressant (n=1); antidepressant dose too low and duration too short (n=1).
Groups:
- Placebo: In this arm, patients will receive placebo for 3 weeks. Placebo identical in appearance to naltrexone will be given twice daily to all patients assigned to placebo.
- Naltrexone: In this arm, patients will receive active naltrexone for 3 weeks. 1 mg of naltrexone will be given twice daily to all patients assigned to active drug.
Period: Overall Study
Arm/Group | Placebo | Naltrexone
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Twenty-one patients were screened, of which twelve patients were admitted into the study, all men and women with major depressive disorder who had relapsed on a pro-dopaminergic antidepressant regimen.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Naltrexone | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (11) | 47 (13) | 45 (12)
Gender [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 3 | 8
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12
Hamilton-D-17 score [Mean (Standard Deviation); unit: units on a scale] — The HAMD-17 contains 17 items covering different depression symptoms. Items are rated on a 0-4 point or 0-2 point scale, where 0 means the symptom is NOT present; higher scores indicate greater symptom severity. Nine items are graded from 0-4 and eight items are rated from 0-2. The highest possible total score on the instrument is 52 and the lowest score is zero. The higher the total score, the greater the depressive severity. As a general guideline, the following total score ranges suggest differing degrees of depression: None = 0-7, Mild = 8-15, Moderate = 16-25, Severe = 26 or greater.
  units on a scale | 23.7 (2.3) | 21.2 (2.0) | 22.4 (2.4)
Hamilton-D-28 score [Mean (Standard Deviation); unit: units on a scale] — The HAMD-28 contains 28 items. Items are rated on a 0-4, 0-3, or 0-2 point scale, where 0 means the symptom is NOT present; higher scores indicate greater symptom severity. Twelve items are graded from 0-4, one from 0-3, and fifteen from 0-2. The highest possible score is 81 and the lowest is 0. higher score means greater severity. Items 18-28 characterize additional symptoms--hypersomnia, hyperphagia, depersonalization, paranoia, and obsessive-compulsive. Overall severity is assessedon the basis of the total score from the first 17 items: None:0-7, Mild:8-15, Moderate:16-25, Severe: >=26.
  units on a scale | 26.3 (2.6) | 26.2 (4.0) | 26.3 (3.2)
MADRS-10 score [Mean (Standard Deviation); unit: units on a scale] — The MADRS-10 contains 10 items, covering different symptoms of depression. Items are equally weighted and scored from 0-6, where 0 indicates that the symptom is NOT present and higher scores indicate greater severity. Thus the highest possible total score on the instrument is 60 and the lowest possible score is zero. The higher the total score, the greater the depressive severity. As a general guideline, the following total score ranges suggest differing degrees of depression: None = 0-6, Mild = 7-19, Moderate = 20-34, Severe = 35 or greater.
  units on a scale | 30.7 (4.3) | 30.4 (4.9) | 30.5 (4.3)
MADRS-15 score [Mean (Standard Deviation); unit: units on a scale] — The MADRS-15 contains 15 items, scored from 0-6, where 0 indicates that the symptom is NOT present and higher scores indicate greater severity. The highest possible score on the instrument is 90 and the lowest 0. The higher the total score, the greater the depressive severity. Items 11-15 characterize additional features of depression including fatigue, psychomotor changes, and hyperphagia and hypersomnia. Overall severity of depression is assessed on the basis of the total score obtained from the first 10 items: None = 0-6, Mild = 7-19, Moderate = 20-34, Severe = 35 or greater.
  units on a scale | 36.7 (4.2) | 36.6 (6.2) | 36.6 (4.9)
Clinical Global Improvement-Severity (CGI-S) score [Mean (Standard Deviation); unit: units on a scale] — The CGI-S score is a one-item scale that measures severity of depression, scored from 1-7, where 1 = no depression is present, 2 = borderline depression, 3 = mild depression, 4 = moderate depression, 5 = marked depression, 6 = severe depression, and 7 = among the most extremely depressed patient. Thus higher scores indicate greater depressive severity.
  units on a scale | 4.3 (0.5) | 4.3 (0.5) | 4.3 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in HAM-D-17 Total Score
Description: Hamilton Depression Scale-17 (HAM-D-17) item. The change in scores depends on the difference between the initial (baseline) score and the final score at the conclusion of the double blind treatment period. There is no formal range of score changes, since they depend on the initial and final score. A negative score represents a lowering in the score from baseline to end (improvement), and a positive score indicates an increase in score from baseline to end (worsening). A zero score would indicate no change. In theory, the maximum drop in score would be from 52 to zero, or -52. A maximum increase would be from 18 (the minimum score required for admission) to 52, or +34.
Time Frame: Change from baseline to week 3
Population: Study completers.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Naltrexone
Number analyzed (Participants) | 6 | 6
units on a scale | -5.8 (5.1) | -9.5 (6.9)

2. Secondary Outcome: Change in HAM-D28 Total Score
Description: Hamilton Depression Scale-28 item. The change in scores depends on the difference between the initial (baseline) score and the final score at the conclusion of the double blind treatment period. There is no formal range of score changes, since they depend on the initial and final score. A negative score represents a lowering in the score from baseline to end (improvement), and a positive score indicates an increase in score from baseline to end (worsening). A zero score would indicate no change. In theory, the maximum drop in score would be from 81 to zero, or -81. A maximum increase would be from 18 (the minimum score required for admission) to 81, or +63.
Time Frame: Change from baseline to week 3
Population: Study subjects who completed the protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Naltrexone
Number analyzed (Participants) | 6 | 6
units on a scale | -6.5 (7.4) | -14.6 (6.7)

3. Secondary Outcome: Change in MADRS-10 Total Score
Description: Montgomery-Asberg Depression Rating Scale- 10 item. The change in scores depends on the difference between the initial (baseline) score and the final score at the conclusion of the double blind treatment period. There is no formal range of score changes, since they depend on the initial and final score. A negative score represents a lowering in the score from baseline to end (improvement), and a positive score indicates an increase in score from baseline to end (worsening). A zero score would indicate no change. In theory, the maximum drop in score would be from 60 to zero, or -60. There is no minimum score on the MADRS-10 required for study entry, since the HAMD-17 was the sole entry criteria. However, a score of 18 on the HAMD17 corresponds to approximately a score of 21 on the MADRS-10. A maximum estimated increase would thus be from 21 to 60, or +39.
Time Frame: Change from baseline to week 3
Population: Study completers.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Naltrexone
Number analyzed (Participants) | 6 | 6
units on a scale | -7.8 (8.5) | -18.2 (5.5)

4. Secondary Outcome: Change in MADRS-15 Total Score
Description: Montgomery-Asberg Depression Rating Scale- 15 item. The change in scores depends on the difference between the initial (baseline) score and the final score at the conclusion of the double blind treatment period. There is no formal range of score changes, since they depend on the initial and final score. A negative score represents a lowering in the score from baseline to end (improvement), and a positive score indicates an increase in score from baseline to end (worsening). A zero score would indicate no change. In theory, the maximum drop in score would be from 90 to zero, or -90. There is no minimum score on the MADRS-15 required for study entry, since the HAMD-17 was the sole entry criteria. However, a score of 18 on the HAMD17 corresponds to approximately a score of 21 on the MADRS-10. A maximum estimated increase would thus be from 21 to 90, or +69.
Time Frame: Change from baseline to week 3
Population: Study completers.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Naltrexone
Number analyzed (Participants) | 6 | 6
units on a scale | -10.7 (10) | -23.4 (6.8)

5. Secondary Outcome: Change in CGI-S Total Score
Description: Clinical Global Improvement-Severity Scale. The CGI-S score is a one-item scale that measures severity of depression, scored from 1-7, where 1 = no depression is present, 2 = borderline depression, 3 = mild depression, 4 = moderate depression, 5 = marked depression, 6 = severe depression, and 7 = among the most extremely depressed patient. Thus higher scores indicate greater depressive severity. The change in CGI-S score can represent a drop from 7 (maximum severity) to 1 (no depression) or -6. There is no minimum CGI-S score required for admission, but a minimum score of 18 on the HAMD17 corresponds to approximately a score of 4 on the CGI-S. Thus a maximum worsening would be from 4 to 7, or +3.
Time Frame: Change from baseline to week 3
Population: Study completers.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Naltrexone
Number analyzed (Participants) | 6 | 6
units on a scale | -0.3 (0.8) | -1.3 (0.8)

6. Secondary Outcome: Final CGI-I Score
Description: Clinical Global Improvement-Improvement Scale. The CGI-I scale is a one item scale that measures overall change in patient's global condition compared to when they were entered into the study. The scale is graded from 1-7, where 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. Thus higher scores indicate greater worsening, and lower scores indicate greater improvement. The lowest possible score (indicating maximum improvement) is 1, and the highest possible score (indicating greatest worsening) is 7.
Time Frame: From baseline to week 3
Population: Study completers.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Naltrexone: In this arm, patients will receive active naltrexone for 3 weeks.1 mg of naltrexone will be given twice daily to all patients assigned to active drug.
Arm/Group | Placebo | Naltrexone
Number analyzed (Participants) | 6 | 6
units on a scale | 3.5 (0.8) | 2.2 (1.2)

7. Secondary Outcome: Response Rate
Description: Response is defined as an improvement in HAM-D-17 score of greater than or equal to 50% compared to baseline score. Response rate is the percent of patients who attain this threshold degree of improvement.
Time Frame: Response rate after 3 weeks
Population: Study completers.
Measure: Count of Participants; unit: Participants
Groups:
- Naltrexone: In this arm, patients will receive low dose naltrexone for three weeks. 1 mg of naltrexone will be given twice daily to all patients assigned to active drug.
Arm/Group | Placebo | Naltrexone
Number analyzed (Participants) | 6 | 6
Participants | 1 | 3
Statistical Analysis 1: Comparison: Placebo vs Naltrexone; Response rates were based on attaining a reduction in the HAM-D-17 scale of 50% or greater compared to baseline. We hypothesized that naltrexone would produce a significantly greater response rate than placebo; Test type: Non-Inferiority or Equivalence — An initial power analysis at the time of protocol development suggested that with 6 patients in each treatment group, we could expect a 79% chance of achieving significance (2-sided p < 0.05) if the true response rate to low-dose naltrexone (LDN) was 80% and the true placebo response rate was 20%; p = 0.55, Chi-squared — Threshold of statistical significance is 0.05; Chi-squared value was 1.5

8. Secondary Outcome: Remission Rate
Description: Remission is defined as a final HAM-D-17 score of 7 or less. Remission rate is the percent of patients who attain this threshold score.
Time Frame: Remission rate at 3 weeks.
Population: Study completers.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naltrexone
Number analyzed (Participants) | 6 | 6
Participants | 0 | 3

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Placebo | Naltrexone
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | Naltrexone (N=6)
Trouble sleeping (Nervous system disorders) | 0 (0) | 2 (2)
Nightmares (Nervous system disorders) | 1 (1) | 0 (0)
Irritable (Psychiatric disorders) | 1 (1) | 0 (0)
Hearing or seeing things (Psychiatric disorders) | 0 (0) | 1 (1)
Numbness or tingling (Nervous system disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Drooling or increased salivation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle cramps or stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tremor or shakiness (Nervous system disorders) | 0 (0) | 1 (1)
Poor coordination or unsteadiness (Nervous system disorders) | 1 (1) | 0 (0)
Trouble catching breath or hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Menstrual irregularities (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Loss of sexual interest (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Problems with sexual arousal (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Delayed or absent orgasm (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Sweating excessively (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fluid retention or swelling (Vascular disorders) | 1 (1) | 0 (0)
Weight gain (General disorders) | 1 (1) | 0 (0)
Strange taste in mouth (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
1) Very small sample. 2) No detailed data about the total number of relapses or recurrences prior to the patients' current regimen. 3) Short double blind treatment period. 4) Focus on antidepressants with dopaminergic activity only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No